CLINICAL TRIAL: NCT01369446
Title: Eeva™ System Study: Noninvasive Recording and Visualization of Individual Embryos Cultured to Blastocyst Stage
Acronym: Eeva
Status: Completed | Type: Observational
Sponsor: Progyny, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TST-1057-p
Record Dates: First submitted 2011-06-07; First posted 2011-06-09 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Infertility
Keywords: In vitro fertilization; Assisted reproduction; Noninvasive imaging of embryos; Time lapse imaging of embryos; Traditional morphological grading of embryos; Prediction of blastocysts
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women undergoing IVF treatment
  Interventions: Device: Eeva System Study

INTERVENTIONS:
Device: Eeva System Study — The Eeva System will image embryos through cleavage and/or blastocyst stage.

SUMMARY:
The purpose of this study is to demonstrate that the Eeva System may be used to identify embryos on Day 2 that are most likely to form blastocysts.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing fresh in vitro fertilization treatment using their own eggs or donor eggs.
* At least 18 years of age.
* Total antral follicle count of at least 12 as measured by ultrasound prior to stimulation.
* Basal FSH < 10 IU.
* At least 8 normally fertilized eggs (2PN.)
* Fertilization using only ejaculated sperm (fresh or frozen) - no surgically removed sperm.
* Willing to comply with study protocol and procedures and able to speak English.

Exclusion Criteria:

* Planned preimplantation genetic diagnosis or preimplantation genetic screening.
* Gestational carriers.
* Use of reinseminated eggs.
* Concurrent participation in another clinical study.
* Previous enrollment in this clinical study.
* History of cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women in the United States who undergo IVF treatment and imaging of their embryos with the Eeva System.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2011-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Eeva System correctly predicts on day 2 those embryos that will reach blastocyst stage at day 5. | Embryos cultured through blastocyst stage (Day 5).
  Imaging data will be manually analyzed to validate parameters previously determined to be predictive of blastocyst formation.

SECONDARY OUTCOMES:
Pregnancy Outcome | Assessed at post embryo transfer day 12-14, post transfer week 5-8, and post transfer week 9-12.
  Chemical pregnancy outcome will be assessed using a serum pregnancy test at post transfer day 12-14. Clinical pregnancy outcome will be assessed using vaginal ultrasound at post transfer week 5-8 and week 9-12. Results will be recorded as positive or negative.

CONTACTS AND LOCATIONS:
Overall Officials: Sheua Shen, MD, ELD, Study Director — Progyny, Inc.
Locations (5):
- United States (5):
  - HRC Fertility, Encino, California
  - Stanford University, Palo Alto, California
  - Pacific Fertility Center, San Francisco, California
  - Fertility Physicians of Northern California, San Jose, California
  - Reproductive Science Center, San Ramon, California

REFERENCES:
- [Background] Wong CC, Loewke KE, Bossert NL, Behr B, De Jonge CJ, Baer TM, Reijo Pera RA. Non-invasive imaging of human embryos before embryonic genome activation predicts development to the blastocyst stage. Nat Biotechnol. 2010 Oct;28(10):1115-21. doi: 10.1038/nbt.1686. Epub 2010 Oct 3. PMID 20890283
- [Derived] Athayde Wirka K, Chen AA, Conaghan J, Ivani K, Gvakharia M, Behr B, Suraj V, Tan L, Shen S. Atypical embryo phenotypes identified by time-lapse microscopy: high prevalence and association with embryo development. Fertil Steril. 2014 Jun;101(6):1637-48.e1-5. doi: 10.1016/j.fertnstert.2014.02.050. Epub 2014 Apr 14. PMID 24726214